CLINICAL TRIAL: NCT05952050
Title: Effect of Different Administration Routes of Dexmedetomidine on Postoperative Delirium in Elderly Patients Undergoing General Anesthesia
Brief Title: Different Administration Routes of Dexmedetomidine on Postoperative Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Intelligent Medical Research Center, Shenzhen United Scheme Technology Co., Ltd. (Industry)
Collaborators: Zhongshan Hospital Of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US2023001
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Dexmedetomidine; Postoperative Delirium; General Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Intravenous dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Different Administration Routes of Dexmedetomidine

SUMMARY:
Intravenous dexmedetomidine has been reported to decrease the occurrence of postoperative delirium (POD) in elderly patients. Nevertheless, some previous studies have indicated that intratracheal dexmedetomidine and intranasal dexmedetomidine are also effective and convenient. The current study aimed to compare the effect of different administration routes of dexmedetomidine on POD in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

Older than 65 years; General anesthesia for more than two hours;

Exclusion Criteria:

-

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of delirium during the first 3 postoperative days | 3 days

SECONDARY OUTCOMES:
The incidence of postoperative sore throat | 3 days
The incidence of sleep quality | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Weitao Chen, Zhongshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided